CLINICAL TRIAL: NCT05880485
Title: A Prospective Study to Evaluate Online Adaptive Radiotherapy in Cervical Cancer With Reduced Margin
Brief Title: Online Adaptive Radiotherapy Cervical Cancer With Reduced Margin for Cervical Cancer
Status: Active, not recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Peking Union Medical College Hospital (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: pumch-ART2
Record Dates: First submitted 2023-04-26; First posted 2023-05-30 (Actual); Last update posted 2024-11-25 (Actual); Status verified 2024-11

CONDITIONS: Uterine Cervical Neoplasm
Keywords: Uterine Cervical Neoplasm; Online Adaptive Radiotherapy
MeSH Terms: conditions — Uterine Cervical Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Online Adaptive Radiotherapy (Experimental): Patients receive online adaptive radiotherapy with 5-10mm PTV margin. The CTV contours of the following areas: gross tumor volume (GTV), cervix (if not already encompassed by the GTV), uterus, parametria, ovaries, vaginal tissue, obturator nodal chain, internal iliac nodal chain, external iliac nodal chain, presacral nodal chain and common iliac nodal chain. The upper border of CTV is at the level of aortic bifurcation. A dose of 50.4Gy is delivered to CTV with online adaptive radiotherapy.
  Interventions: Radiation: online adaptive radiotherapy

INTERVENTIONS:
Radiation: online adaptive radiotherapy — PTV with 5-10 margins covers CTV

SUMMARY:
Online adaptive radiotherapy (oART) has demonstrated to be feasible to reduce planning target volume (PTV) margins for cervical cancer. To explore the value of reduced margins in oART for cervical cancer, we conducted a prospective clinical trial to determine the clinical efficacy and toxicity of reduced margins.

DETAILED DESCRIPTION:
This is an investigator-initiated efficacious, single-center, open-label clinical trial study. This study hypothesizes that the use of reduced PTV margins in oART for cervical cancer could decrease toxicity and achieve more accurate dosimetric coverage. A dose of 50.4 Gy is delivered to clinical target volume (CTV) with reduced margin oART. Patients receive cisplatin based concurrent chemotherapy. The primary endpoint is acute toxicity.

ELIGIBILITY:
Inclusion Criteria:

1. Patients must be informed of the investigational nature of this study and give written informed consent before treatment.
2. Age ≥18 years and ≤ 75 years.
3. Patients with newly histologically confirmed cervical cancer, including squamous cell carcinoma, adenocarcinoma and adenosquamous carcinoma, et al.
4. No evidence of para-aortic metastatic lymph nodes (MLNs) and inguinal lymph nodes on CT, MRI or positron emission tomograph (PET)/CT.
5. No contraindications to CT scanning.
6. No evidence of distant metastasis (FIGO stage IVB).
7. Adequate marrow: neutrophile granulocyte count ≥1.5*10^9/L, hemoglobin ≥ 80 g/L, platelet count ≥100*10^9/L.
8. Normal liver and kidney function: Creatinine (Cr) < 1.5 mg/dl, Alanine Aminotransferase (ALT), Aspartate Aminotransferase (AST) < 2*upper limit of normal (ULN).

Exclusion Criteria:

1. With common iliac MLNs.
2. Tumor extended to the lower third of the vagina.
3. Tumor spread to mucosa of the bladder or rectum.
4. Prior surgery (including pelvic or para-aortic lymph nodes resection, except for tumor biopsy), radiotherapy or chemotherapy to primary tumor or nodes.
5. Prior malignancy.
6. History of previous radiotherapy to the abdomen or pelvis.
7. Pregnancy or lactation.
8. Active inflammatory bowel disease, or history of severe stomach or duodenal ulcer.
9. Active infection with fever.
10. Patients with unacceptable risk that intracavitary brachytherapy can not be conducted.
11. Any severe disease which may bring unacceptable risk or affect the compliance of the trial, for example, unstable cardiac disease requiring treatment, renal disease, chronic hepatitis, diabetes with poor control, and emotional disturbance.

Ages: 18 Years to 75 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2023-02-02 (Actual); Primary Completion 2023-11-06 (Actual); Study Completion 2025-11 (Estimated)

PRIMARY OUTCOMES:
Patient-reported acute toxicity | From the start of treatment to 3 months after treatment
  Patient-reported acute toxicity evaluated with European Organization for Research and Treatment of Cancer Quality of Life C30 (EORTC QLQ-C30) 3.0 questionnaire
Physician-reported acute toxicity | From the start of treatment to 3 months after treatment
  Physician-reported acute toxicity evaluated with Common Terminology Criteria for Adverse Events (CTCAE) 5.0

SECONDARY OUTCOMES:
Late toxicity evaluated with Radiation Therapy Oncology Group (RTOG)/EORTC late radiation morbidity scoring scheme | 2-year
  Evaluated with Radiation Therapy Oncology Group (RTOG)/EORTC late radiation morbidity scoring scheme
The irradiated doses of organs at risk | Through study completion, an average of eight month
  The organs at risk includes bladder, rectum, bone marrow, femur head left, femur head right and bowel that may be irradiated near the target volume
The dose coverage of target volume as assessed by planing tumor volume V100% | Through study completion, an average of eight month
  Planing tumor volume V100%, defined as the planing tumor volume receiving at least 100% of the prescribed dose (V100%), is used to evaluate the dose coverage of target volume.
Target volume contouring accuracy | Through study completion, an average of eight month
  For every target in each fraction, the evaluation of accuracy for target contouring are categorized as follow: no edits, minor edits, moderate edits, major edits and not applicable.
Response evaluation evaluated with RECIST 1.1 | One month after treatment
  Evaluated with RECIST 1.1
Movement of the uterus during per radiotherapy fractions | Through study completion, an average of eight month
  The pre- and post-treatment CBCT scans will be obtained during per treatment. The uterus intra-fractional motion were evaluated by comparison of uterus centroid from pre-treatment CBCT and uterus centroid from post-treatment images.
Movement of the cervix during per radiotherapy fractions | Through study completion, an average of eight month
  The pre- and post-treatment CBCT scans will be obtained during per treatment. The cervix intra-fractional motion were evaluated by comparison of cervix centroid from pre-treatment CBCT and cervix centroid from post-treatment images.
Progression-free survival | 2-year
  Progression-free survival is defined as the time from randomization to disease progression or death from any cause, whichever is first.
Personalized margin for cervical cancer | Six month after treatment
  Pre- and post-treatment images are uploaded to the online adaptive radiotherapy simulator to re-delineate the target volume and determine the personalized margin range.

CONTACTS AND LOCATIONS:
Overall Officials: Fuquan Zhang, M.D., Study Chair — Peking Union Medical College Hospital
Locations (1):
- Peking Union Medical College Hospital, Beijing, Beijing Municipality, China

REFERENCES:
- [Background] de Jong R, Visser J, van Wieringen N, Wiersma J, Geijsen D, Bel A. Feasibility of Conebeam CT-based online adaptive radiotherapy for neoadjuvant treatment of rectal cancer. Radiat Oncol. 2021 Jul 23;16(1):136. doi: 10.1186/s13014-021-01866-7. PMID 34301300
- [Result] Yen A, Choi B, Inam E, Yeh A, Lin MH, Park C, Hrycushko B, Nwachukwu C, Albuquerque K. Spare the Bowel, Don't Spoil the Target: Optimal Margin Assessment for Online Cone Beam Adaptive Radiation Therapy (OnC-ART) of the Cervix. Pract Radiat Oncol. 2023 Mar-Apr;13(2):e176-e183. doi: 10.1016/j.prro.2022.10.009. Epub 2022 Nov 7. PMID 36356834